CLINICAL TRIAL: NCT04677023
Title: Clinical Evaluation of Organically Modified Ceramic Resin Composite Versus Conventional Bulkfill Resin Composite in Proximal Compound Posterior Restorations: Randomized Clinical
Brief Title: Evaluation of Organically Modified Ceramic Resin Composite Versus Bulkfill Resin in Proximal Posterior Cavities
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, safinaz hussien fahmy hassan, principle investegator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 88960
Record Dates: First submitted 2020-09-15; First posted 2020-12-21 (Actual); Last update posted 2020-12-23 (Actual); Status verified 2020-12

CONDITIONS: Proximal Caries

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Admira fusion X--tra® bulk (Other): The special ORMOCER® compound molecules in Admira Fusion x-tra reduce the volume shrinkage to an extremely low level (1.25 % by volume) in conjunction with very low shrinkage stress (3.87 MPa). Admira Fusion x-tra is the bulk fill version of Admira Fusion. This means that this restorative material can be applied in layers of up to 4 mm and then reliably cured. This makes placing posterior restorations particularly quick and economical. The universal shade U further simplifies handling, as it provides aesthetic results by adapting, chameleon-like, to the surrounding dental substance
  Interventions: Other: Admira fusion X--tra® bulk
- GrandioSO x-tra® bulk (Other): a nano-hybrid composite which is in a class of its own. It is distinguished by outstanding handling and excellent physical properties, modelled on the natural tooth.its the packable bulk fill material for the highest standards in durability and aesthetics.GrandioSO x-tra has outstanding surface hardness, at 223 MHV, which is closer to natural tooth enamel, compared with other bulk fill composites. Because of this, GrandioSO x-tra ensures restorations which are abrasionresistant and dimensionally stable over the long term. In addition to the surface hardness, reliable curing is very important when larger increments are used. Here as well, GrandioSO x-tra achieves an outstanding result and, at the 219 MHV measured at a depth of 4 mm, it even significantly exceeds the values measured for other bulk fill composites at the surface.
  Interventions: Other: GrandioSO x-tra® bulk

INTERVENTIONS:
Other: GrandioSO x-tra® bulk — The prepared cavities will be restored with GrandioSO X-tra (VOCO, Cuxhaven, Germany) in layers that are a maximum of 4 mm thick then cured for 20 seconds using using Elipar™️ S10 LED curing light (3M ESPE, St Paul, MN, USA) with light intensity of 1200 mW/cm2.
  Arms: GrandioSO x-tra® bulk
Other: Admira fusion X--tra® bulk — he prepared cavities will be restored with Admira fusion X-tra®️ bulk (VOCO, Cuxhaven, Germany) in layers that are a maximum of 4 mm thick then cured for 20 seconds using usingElipar™️ S10 LED curing light (3M ESPE, St Paul, MN, USA) with light intensity of 1200 mW/cm2.
  Arms: Admira fusion X--tra® bulk

SUMMARY:
In patients with compound posterior proximal cavities, will the use of organically modified ceramic resin composite restorative material have similar clinical performance to conventional bulk fill resin composite, evaluation of restorations will be done at baseline,six and twelve months using World Dental Federation FDI criteria.

DETAILED DESCRIPTION:
The study will be conducted in the clinic of Conservative Dentistry Department, Faculty of Dentistry, Cairo University; the operator in charge Safinaz Hussien ,The subjects fulfilling the eligibility criteria of the trial will be selected from the regular attendees at the clinic of Conservative Dentistry Department, Faculty of Dentistry, Cairo University.Patient examination will be done including medical history, dental history, extra-oral examination and intra-oral examination. A periapical radiograph will be taken prior to restorative procedures to assess the degree of approximation of caries to pulp, intactness of lamina dura and/or presence of any periapical radiolucency to exclude the case.The field of operation will be isolated with the application of a rubber dam if possible. Otherwise, cotton rolls and the saliva ejector will be used for moisture control. For cavity preparation, local anesthetic (Mepecaine-L, Alexandria Company, Egypt) solution will be administrated to control patient discomfort during the procedure.The cavities will be prepared by using cylindrical #314 (Komet®, Germany) in a high speed handpiece (Sirona, Germany) rotating at high speed with copious coolant. Remaining soft caries -if present- will be removed using sharp excavator (Maillefer, Dentsuply, Switzerland).After the cavity preparation is finished, it will be thoroughly air-water cleaned. The bonding system; FuturabondU(Voco, Germany) will be applied according to the following instructions recommended by the manufacturer: Futurabond M+ will be applied to prepared tooth structure and cured for 20 seconds using Elipar™ S10 LED curing light (3M ESPE, St Paul, MN, USA) with light intensity of 1200 mW/cm2. The prepared cavities will be restored with Admira fusion X--tra® bulk (VOCO, Cuxhaven in layers that are a maximum of 4 mm thick then cured for 20 seconds using usingElipar™ S10 LED curing light (3M ESPE, St Paul, MN, USA) with light intensity of 1200 mW/cm2. and for the control group cavities will be restored with GrandioSO x-tra(VOCO, Cuxhaven) in layers that are a maximum of 4 mm thick then cured for 20 seconds using usingElipar™ S10 LED curing light (3M ESPE, St Paul, MN, USA) with light intensity of 1200 mW/cm2.

ELIGIBILITY:
Inclusion Criteria:

* Patients aging ≥18 years.
* Patients with a high level of oral hygiene.
* Patients having at least 1or 2 posterior teeth in occlusion.
* Patients with good likelihood of recall availability.

Tooth inclusion:

* Permanent premolars or molars.
* Moderate to deep compound class II cavities.
* Primary carious lesions.
* Vital with positive reaction to cold thermal stimulus.
* Well-formed and fully-erupted in normal functional occlusion with natural antagonist and adjacent teeth.

Exclusion Criteria:

* Participants with general/systemic illness.
* Pregnant or lactating females.
* Concomitant participation in another research study.
* Inability to comply with study procedures.
* Heavy bruxism habits.
* Last experience with allergic reactions against any components of the used materials.
* Patients receiving orthodontic treatment.

Tooth exclusion:

* Teeth with clinical symptoms of pulpitis such as spontaneous pain or sensitivity to pressure.
* Non-vital teeth.
* Secondary carious lesions.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Estimated)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-02-01 (Estimated)

PRIMARY OUTCOMES:
Fracture | 24 months
  Fracture of material visually inspected and evaluated using FDI probe and then classified accordingly
  1. clinically excellent/very good: No fractures /cracks.
  2. Clinically good: Small hairline crack.
  3. Clinically sufficient /satisfactory(minor shortcomings, no unacceptable effects but not adjustable w/or damage to the tooth):Two or more or larger hairline cracks and/or material chipfracture no affecting the marginal integrity or approximal contact.
  4. Clinically unsatisfactory /(but reparable):Material chip fractures which damage marginal quality or Bulk fractures with partial loss(less than half of the restoration). ditching or marginal fractures.
  5. Clinically poor (replacement necessary): (Partial or complete) loss of restoration or multiple fractures.

SECONDARY OUTCOMES:
color match | 24 months
  Esthetic visually inspected and evaluated using FDI probe and then classified
  1. clinically excellent/very good Luster comparable to enamel,& , no difference in shade
  2. Clinically good Slightly dull, & minor shade deviation
  3. Clinically sufficient /satisfactory. Dull surface & distinct shade deviation
  4. Clinically unsatisfactory /(but reparable) Rough surface, & localized shade deviation that can be repaired
  5. Clinically poor (replacement necessary): Very rough & un acceptable shade need replacement

OTHER OUTCOMES:
secondary caries | 24 months
  Biological properties: visually inspected and evaluated using FDI probe and then classified accordingly
  1. Clinically excellent / very good no caries
  2. Clinically good small & localized
  3. Clinically sufficient /satisfactory large area of demineralization
  4. Clinically unsatisfactory (but reparable) caries with cavitation
  5. Clinically poor (replacement necessary) Deep caries or exposed dentine

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: expecting to have all the data by October 2022